CLINICAL TRIAL: NCT07190989
Title: Inter-individual Variability of Sleep Outcome Measures in Response to Nutritional Blend Supplementation: a Replicate Crossover Trial
Brief Title: A Replicate Crossover Trial on Nutritional Supplementation in Association Football (Soccer)
Acronym: AANOF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aspire Academy (Other Government)
Responsible Party: Principal Investigator, Lorenzo Lolli, Principal Investigator, Aspire Academy
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: F202501089
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: actigraphy; ergogenic dietary supplements; replicate crossover; individual variability
MeSH Terms: interventions — Dietary Supplements; maltodextrin

STUDY DESIGN:
Intervention Model Description: Replicate crossover trial design involving repeated administration of both supplementation and placebo conditions over 2 cycles involving 2 administrations of supplementation and 2 administrations of placebo in a randomized order (four periods in total). Additional information and details are available in Senn (2016).
  References
  Senn S. Mastering variation: variance components and personalised medicine. Stat Med. 2016;35(7):966-977.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation (Experimental): In the absence of established target difference and design-specific variance values relevant to each primary outcome measure considered in this study, and in keeping with procedures adopted to sample size justification in previous research adopting a replicate crossover design (Gonzalez et al., 2024), a minimum sample size of 12 participants would translate to a one-tailed between-cycle correlation of 0.5, with a 90% confidence interval for this correlation ranging from 0.00 to 0.80, assuming a null and a negative correlation would suggest non-rejection of the null hypothesis (r ≤ 0). The treatment administration will involve a nutritional blend consisting of a mixed juice containing 15000 mg cherry juice concentrate, 220 mg cherry extract, 250 mg cocoa extract, 200 mg of tryptophan, 100 mg of L-5-Hydroxytryptophan, 3000 mg of glycine, 300 mg of magnesium, 200 mg of Theanine manufactured by Science in Sport (https://sport.wetestyoutrust.com/supplement-search/science-sport/rest-juice).
  Interventions: Dietary Supplement: Nutritional Supplement
- Placebo (Placebo Comparator): In the absence of established target difference and design-specific variance values relevant to each primary outcome measure considered in this study, and in keeping with procedures adopted to sample size justification in previous research adopting a replicate crossover design (Gonzalez et al., 2024), a minimum sample size of 12 participants would translate to a one-tailed between-cycle correlation of 0.5, with a 90% confidence interval for this correlation ranging from 0.00 to 0.80, assuming a null and a negative correlation would suggest non-rejection of the null hypothesis (r ≤ 0). The placebo treatment will involve a 40g dual-source carbohydrate gel, having a 1:0.8 ratio of maltodextrin and fructose, as an alternative supplementation known for having trivial effects on sleep-related outcome measures (https://sport.wetestyoutrust.com/supplement-search/science-sport/beta-fuel-dual-source-energy-gel-beta-fuel-maltodextrin-fructose).
  Interventions: Dietary Supplement: Maltodextrin (Placebo)

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — A mixed juice containing 15000 mg cherry juice concentrate, 220 mg cherry extract, 250 mg cocoa extract, 200 mg of tryptophan, 100 mg of L-5-Hydroxytryptophan, 3000 mg of glycine, 300 mg of magnesium, 200 mg of theanine manufactured by Science in Sport (https://sport.wetestyoutrust.com/supplement-search/science-sport/rest-juice).
  Arms: Supplementation
Dietary Supplement: Maltodextrin (Placebo) — A 40g dual-source carbohydrate gel, having a 1:0.8 ratio of maltodextrin and fructose manufactured by Science in Sport (https://sport.wetestyoutrust.com/supplement-search/science-sport/beta-fuel-dual-source-energy-gel-beta-fuel-maltodextrin-fructose).
  Arms: Placebo

SUMMARY:
Problems of sleep disorders and disruption are common particularly in Arab populations, and sleep insufficiency hinders the pursuit of high performance and optimal recovery following training and competition. Adequate investigation and personalization of dietary interventions to enhance sleep and recovery requires employing suitable methods of experimentation that involves repeated administration of treatment and placebo conditions, following a replicate crossover trial design, for derivation of athlete by dietary treatment interaction to inform decisions of supplementation dosing personalization embedded into routine service provision. Nevertheless, no study in sports performance explored this and other issues following adequate methodology and research design requirements. Accordingly, the project seeks to investigate the main effects and whether inter-individual variability exists in free-living objective sleep and recovery responses to novel nutritional blend supplementation in the form of a mixed juice (15000 mg cherry juice concentrate, 220 mg cherry extract, 250 mg cocoa extract, 200 mg of tryptophan, 100 mg of L-5-Hydroxytryptophan, 3000 mg of glycine, 300 mg of magnesium, 200 mg of theanine) adopting a replicate crossover design.

DETAILED DESCRIPTION:
Background information & study rationale: A number of investigations explored the effects nutritional supplements on proxy measures of sleep and recovery. Notably, different studies examined the properties of high glycemic index carbohydrates, tryptophan, tart cherries, glycine, magnesium, and L-theanine predominantly in isolation in sample of participants from general populations with and without sleep disorders. However, none of these studies involved elite athletes nor assessed the effects of and potential for personalizing nutritional supplementation according to evidence from appropriately designed experimental investigations involving the repeated administration of supplementation and placebo conditions adopting a replicate crossover trial design. With this in mind, and for the first time, the project seeks to quantify the magnitude of inter-individual variability in the effects of a novel nutritional blend supplementation in the form of a mixed juice (15000 mg cherry juice concentrate, 220 mg cherry extract, 250 mg cocoa extract, 200 mg of tryptophan, 100 mg of L-5-Hydroxytryptophan, 3000 mg of glycine, 300 mg of magnesium, 200 mg of theanine - https://sport.wetestyoutrust.com/supplement-search/science-sport/rest-juice) on proxy measures of recovery and sleep using a replicate crossover design. The project seeks to examine the consistency of these responses on repeated occasions. We hypothesize that there is 'true' inter-individual variability (i.e., exceeding random within-subject variability) in the effects of nutritional blend supplementation on actigraphy-based sleep outcome measures and proxies of recovery, and that these responses would be consistent on two occasions. Adequate sleep and recovery are pivotal to promote optimal preparation training and competition as well as foster high performance in elite sport (Fox et al., 2020). Importantly, continuous unperturbed sleep represents a physiological necessity to preserve normal cognitive and neurobehavioral functions (Maquet 2001; Van Someren et al. 2015; Logan and McClung 2019; Walsh et al. 2020). Nevertheless, youth athletes are vulnerable to sleep disorders that generally involve short durations inconsistent with health recommendations due to lifestyle factors, social commitments (e.g., school), coupled with the demands of training and competition (Fox et al. 2020). In this context, Muslim from general and athletic populations are particularly prone to issues of sleep disorders and schedule congestion throughout different seasons of the Gregorian year. Outcomes from a 14-day surveillance period from Aspire Academy youth football players (Lolli et al., 2021) were consistent with this line of evidence that highlighted children, adolescents, and young adults from Qatar do not meet the age-specific sleep recommendations (i.e., 8 hr to 9 hr of sleep per night). Furthermore, recent findings highlighted how the observance of the holy month of Ramadan exacerbated such issues in Aspire Academy student-athletes, with an average 4.2 hr (95% confidence interval, 3.6 to 4.7 hr) in the first block of night sleep immediately after Ramadan onset (Lolli et al., 2024a). From a clinical standpoint, sleep insufficiency issues can potentially disrupt a student-athlete's biological clock via desynchronisation of its key modulators, such as leptin, adiponectin and ghrelin, involved in appetite regulation and energy expenditure (Knutson et al., 2007). A recent randomized, controlled, crossover, 21-day inpatient study revealed experimental sleep restriction (i.e., 4 hr of night sleep) in free access to food conditions (i.e. ad libitum) caused increased energy intake with no changes in energy expenditure, leading to significant weight gain (Covassin et al., 2022). On the other hand, inconsistent eating habits might impair energy balance that, as a consequence, can offset and be detrimental to the youth athlete development process (Mountjoy et al., 2018). To address such issues, while also considering the number of narrative review and consensus statements, a number of studies in the literature examined various nutritional ingredients with proposed recovery and sleep enhancing qualities involving high glycemic index carbohydrates, tryptophan, tart cherries, glycine, magnesium, and L-theanine (Langan-Evans et al., 2023) yet without adopting appropriate research designs to explore the main effects and potential for personalization based on the assessment of interindividual differences in responses explored in elite athletes. Identification of meaningful inter-individual differences in response to nutritional interventions can be challenging. Notably, with conventional parallel-arm or crossover trials, it is not possible to determine whether any apparent difference between participants in the changes from pre- to post-intervention are due to genuine treatment response heterogeneity or are a consequence of random within-subject variability and/or measurement error (Senn 2016). Without repeated administration of trials, a typical crossover design does not allow formal estimation of variance attributable to participant-by-treatment interaction (Atkinson and Batterham, 2015; Senn 2019). Only with knowledge about this interaction can treatment response heterogeneity be quantified properly. As a form of n-of-1 trial, a replicate crossover trial constitutes a pragmatic research design for quantifying treatment response heterogeneity (Atkinson and Batterham, 2015; Senn et al., 2011; Senn 2016). This research design involves repeated administration of the intervention and control/placebo arms of a trial protocol in randomized order on at least two occasions. This design allows a principled estimation of various components of variation to examine whether genuine supplementation response heterogeneity can be distinguished from random within-subject variability for researchers to arrive at appropriate conclusions on the presence and consistency of inter-individual differences in the supplementation administration responses (Senn et al., 2011). Nevertheless, these aspects remain unexplored in the sports performance literature the modern Arab paediatric population from the State of Qatar. Notably, no study in the sports performance literature adopted a replicate crossover design to examine the possibility of personalized recommendations for dietary supplementation for optimal post-training and post-competition recovery management.

Study goals and objectives: To investigate the main effects and whether inter-individual variability exists in free-living objective sleep and subjective training load responses to novel nutritional blend supplementation in the form of a mixed juice (15000 mg cherry juice concentrate, 220 mg cherry extract, 250 mg cocoa extract, 200 mg of tryptophan, 100 mg of L-5-Hydroxytryptophan, 3000 mg of glycine, 300 mg of magnesium, 200 mg of theanine) adopting a replicate crossover design for exploring whether it may work in youth athletes and the potential for supplement administration personalization.

Study Design and Research Population: Considering the nature of a replicate crossover trial being an alternative form of n-of-1 trial in which each participant will represent a distinct trial and will act as his own control (Senn 2019), the present investigation will aim to assess the effects of nutritional supplementation embedded into routine service provision settings. Accordingly, the target sample will involve youth football players (target age range: 13 to 17 years) that will follow a period of preparation in the lead to the FIFA U-17 World Cup.

Description of subjects: Considering the nature of a replicate crossover trial being an alternative form of n-of-1 trial in which each participant will represent a distinct trial and will act as his own control (Senn 2019), the present investigation will aim to assess the effects of nutritional supplementation in routine service provision settings. Accordingly, the target sample will involve youth football players (target age range: 13 to 17 years) that will follow a period of preparation in the lead to the FIFA U-17 World Cup. In the absence of established target difference (Cook et al., 2018) and design-specific variance (Senn, 2019) values relevant to each primary outcome measure considered in this study, and in keeping with procedures adopted to sample size justification in previous research adopting a replicate crossover design (Gonzalez et al., 2024), a minimum sample size of 12 participants would translate to a one-tailed between-cycle correlation of 0.5, with a 90% confidence interval for this correlation ranging from 0.00 to 0.80, assuming a null and a negative correlation would suggest non-rejection of the null hypothesis (r ≤ 0).

Methodology: The study methods definition will follow the recent guidance (Chatters et al., 2024) and the Consolidated Standards of Reporting Trials (CONSORT) 2010 statement extended to randomized (replicate) crossover trials (Dwan et al., 2019). The relevant checklist (Dwan et al., 2019) for the design and conduct of the study will be completed accordingly. Using a replicate crossover design (Senn 2016), participants will complete two identical supplementation and two identical placebo l trials in a randomized order separated by at least four days. The randomization sequence for the four experimental trials will be conducted using the PLAN procedure available in SAS (Deng & Graz, 2002). The supplement treatment will involve administering a nutritional blend consisting of a mixed juice containing 15000 mg cherry juice concentrate, 220 mg cherry extract, 250 mg cocoa extract, 200 mg of tryptophan, 100 mg of L-5-Hydroxytryptophan, 3000 mg of glycine, 300 mg of magnesium, 200 mg of Theanine sought to be manufactured by Science in Sport (https://sport.wetestyoutrust.com/supplement-search/science-sport/rest-juice) and within safety limits for administration in children and adolescents (Barrett et al., 2013; Bruni et al., 2004; Cynober et al., 2016; Elango, 2023; Fernstrom, 2012; Garlick, 2004; Institute of Medicine Standing Committee on the Scientific Evaluation of Dietary Reference, 1997; Lyon et al., 2011; Merry and Ristow, 2016; Rose et al., 1965). The placebo will involve a 40-g dual-source carbohydrate gel, having a 1:0.8 ratio of maltodextrin and fructose, as an alternative supplementation known for having trivial effects on sleep-related outcome measures (St-Onge et al., 2016). Both the supplement and the placebo will be administered in a random order across 2-night period for each respective main trial separated 5-day washout periods to mitigate carryover effects between trial periods and cycles consistent with the squad microcyle planning. The supplement and placebo administration will mimic a post-match recovery context, with both treatment conditions being administered within 1-hour post-training and coinciding with dinner time. Both the participant and the performance nutritionist administering the supplementation will be blinded to its administration and treatment episode allocation. The washout diet will involve an "eat as usual" protocol consistent with recommendations by Aspire Academy sports nutrition recommendations refraining from any caffeine and nicotine consumption. Participants will be required to undertake a food diary using the remote food photography method as previously utilised in adolescent male football players (Hannon et al., 2021). In brief, participants will be instructed on how to capture photographs at 45 degrees and 90 degrees angles before and after each eating and/or drinking occasion, which will be recorded and time stamped via WhatsApp (WhatsApp Inc., Mountain View, CA) as previously described (Hannon et al., 2021). These data will then be assessed by two accredited sports nutrition practitioners using dietary analysis software to establish daily energy and macronutrients values (Nutritics V5, Nutritics Ltd, Swords, Co. Dublin, Ireland). Parents of the participants will be fully informed regarding the aim of the study, however, the participants will be informed that the study's aim is to measure the effect of two supplemental treatments on physical performance outcomes. The intention of this deception blinding is to make participants unaware of the true aim of the study. A run-in period one week prior to formal trial initiation is considered to determine tolerability and assess potential compliance with study regimens (Shamseer et al., 2015), although no major risks are foreseen. Importantly, the adoption of replicate crossover trial design allows to maximize resources by minimizing participant recruitment requirements of parallel-arm trials requiring a larger pool of participants (Nikles et al., 2011). In a replicate crossover trial, each participant represents a distinct trial and will act as his own control (Senn 2019). Aggregation of each trial will be relevant to derive population- and individual-based estimates regarding supplementation effectiveness (Zucker et al., 1997).

Description of the drug/device/vaccine/dietary intake that is being tested or in social sciences for example providing training or information to groups of individuals: The supplement treatment will involve administering a nutritional blend of natural ingredients consisting of a mixed juice containing 15000 mg cherry juice concentrate, 220 mg cherry extract, 250 mg cocoa extract, 200 mg of tryptophan, 100 mg of L-5-Hydroxytryptophan, 3000 mg of glycine, 300 mg of magnesium, 200 mg of theanine sought to be manufactured by Science in Sport (https://sport.wetestyoutrust.com/supplement-search/science-sport/rest-juice) and within safety limits for administration in children and adolescents (Barrett et al., 2013; Bruni et al., 2004; Cynober et al., 2016; Elango, 2023; Fernstrom, 2012; Garlick, 2004; Lyon et al., 2011; Merry and Ristow, 2016; Rose et al., 1965). The placebo will involve a 40-g dual-source carbohydrate gel, having a 1:0.8 ratio of maltodextrin and fructose, as an alternative supplementation known for having trivial effects on sleep-related outcome measures (St-Onge et al., 2016). Supplementation may elicit potential gastrointestinal discomfort and presents minimal risks that, if occur, will involve the student-athlete withdrawing from the study. A run-in period one week prior to formal trial initiationmay be considered to determine tolerability and assess potential compliance with study regimens (Shamseer et al., 2015), although no major risks are foreseen. Nevertheless, the length of our protocol washout periods is deemed adequate to mitigate any unforeseeable issue due to potential side effects. Both active supplementation (https://sport.wetestyoutrust.com/supplement-search/science-sport/rest-juice) and placebo (https://sport.wetestyoutrust.com/supplement-search/science-sport/beta-fuel-dual-source-energy-gel-beta-fuel-maltodextrin-fructose) are Informed Sport Tested since commercially available. Informed Sport is the world's leading testing and certification program for brands producing sports and nutritional supplements. Designed for elite sport, it protects athletes from inadvertent doping caused by supplements contaminated with banned substances.

Procedures: Time asleep, defined as 'the actual time that a person spends asleep excluding non- sleep-related activities in bed', will represent the primary outcome measure in this investigation (Reed and Sacco 2016). Secondary outcome measures were ratings of perceived exertion (RPE; au) on the CR-100 scale and a proxy measure of high-intensity activity determined as high-speed running distance in meters (Borg 1998; Di Salvo et al. 2009). Time in bed and wake-after-sleep-onset represented other secondary outcome measures (Reed and Sacco 2016). Study participants will wear an ActiGraph GT9X Link (ActiGraph, Pensacola, FL, USA) activity monitor set for date of birth, stature, body mass, and non-dominant wrist. Devices will track all activities during the surveillance period except involvement in training and official matches only. The ActiGraph GT9X Link monitors (35mm×35mm×100mm, and a weight of 14 g) will be configured as per the manufacturer recommendations, with the Cole-Kripke sleep scoring algorithm used to analyze the data and the Tudor-Locke algorithm (Tudor-Locke et al. 2014) set as default for automated sleep period detection (Cole et al. 1992; Quante et al. 2018). Student-athletes will rate the global intensity (RPE) of all sessions using level-anchored semi-ratio Borg CR-100® scale (Borg 1998). Running distances will be monitored during all training sessions with 10-Hz global positioning system (GPS; Fitogether). In line with procedures outlined by Short et al., 2017, participants will be provided with sleep diary for completion during the selected observational time. The purpose of using a sleep diary intends to gather the following information: time someone went to bed; time someone thought fell asleep; time someone woke up (Short et al., 2017). A run-in period one week prior to formal trial initiation will be considered to determine tolerability and assess potential compliance with study regimens (Shamseer et al., 2015), although no major risks are foreseen. The randomization sequence for the four experimental trials will be conducted using the PLAN procedure available in SAS (Deng & Graz, 2002). Both the participant and the performance nutritionist administering the supplementation will be blinded to its administration and treatment episode allocation.

Procedures for analysis and Interpretation of Data: The statistical analysis framework involves a four-step approach in line with existing research (Senn et al., 2011; Senn 2016; Goltz et al., 2018; Goltz et al., 2019; Shen et al., 2024) and more recent advances (Senn 2024) for appropriate examination of continuous data from a replicate crossover experiment. Response pairs will be formulated by calculating the placebo-adjusted treatment effect for the first supplementation and placebo pair in each participants' sequence (response 1; supplementation 1 minus placebo 1) along with the second supplementation and placebo pair (response 2; supplementation 2 minus placebo 2). The first and second replicates will be calculated as the difference between the supplementation and placebo trial pre-to-post change scores in two comparisons:

1. The immediate impact of supplementation minus placebo on the first administration night;
2. The immediate impact of supplementation minus placebo for the outcome average over the two administration nights as a summary measure (Senn, 2000; Yang et al., 2025).

First, estimation of Pearson's product moment correlation coefficients between the two replicates of the supplementation and placebo differences for each sleep outcome (Senn 2016) is relevant to explore the consistency of the supplementation effect between the replicate trials, with thresholds of 0.1, 0.3 and 0.5 indicating small, moderate and large coefficients, respectively. Second, a naïve estimate (estimate 1) of the true (placebo-adjusted) individual differences SD will be determined by calculating the difference in SDs of the pre-to-post change between the supplementation and placebo trials (Atkinson and Batterham, 2015; Atkinson et al., 2019). These calculations utilise the appropriate equation for pooling SDs across the two replicates of the supplementation and placebo trials. A positive SDIR indicates greater heterogeneity in the supplementation response compared to any random within-subject variability. Third, separate within-participant linear mixed modelling will conducted in SAS OnDemand for Academics for each outcome to derive the participant-by-trial interaction which models trial, period (trial sequence) and the period-by-trial interaction as fixed effects, whereas participant and the participant-by-trial interaction will be modelled as random effects. Estimate 2 of the true individual differences SD will be derived from the participant-by-trial interaction term. Standard residual diagnostics will be performed to assess the adequacy and stability of the modelled covariance parameter estimates and a sensitivity analysis will be conducted excluding outliers that were > 3 times higher or lower than the sample SD. Fourth, a sample estimate of within-subjects variance will be calculated and converted it to a standard error using appropriate degrees of freedom given the completed cycles to derive per participant replicate-averaged treatment effects (Senn 2024). A random-effects meta-analysis with Hartung-Knapp adjustment (IntHout et al., 2014) will summarise individual-participant replicate-averaged treatment effects and respective sampling errors (Senn 2024) conducted using the metagen() function. The restricted maximum-likelihood estimation method will determine the tau-statistic (τ) value describing the between-participant replicate-averaged treatment effect response variability across the distribution of true supplementation-related effects (Langan et al., 2019; Veroniki et al., 2016) The uncertainty surrounding the point τ-statistic estimate was described using 95% CI derived using the generalised Q-statistic method (Viechtbauer 2007) Weighted raw replicate-averaged treatment effects will be reported as descriptive statistics alongside the respective 95% prediction interval illustrating the range for the distribution of true mean differences expected for 95% of similar trials (Borenstein 2024; IntHout et al., 2016) Meta-analyses will be conducted in R (version 3.6.3, R Foundation for Statistical Computing). Mean differences and correlation coefficients will be reported with their corresponding 95% confidence intervals (CI). Accordingly, the phenomenon of statistical shrinkage of treatment effects toward the sample-level mean by deriving best linear unbiased predictor, or shrunk, estimates using the blup() function following random effects meta-analysis modelling using the metafor package (Senn, 2024). Visual inspection of unadjusted (or naïve) estimates (x-axis) against shrunk estimates (y-axis) informed judgements relevant to interpreting the clinical meaningfulness of the estimated response heterogeneity. A minimal clinical important difference (MCID) of ± 30 minutes will inform interpretations for time asleep and total time in bed variables. These values are in line with proposed thresholds defining the acceptable difference in sleep outcomes between actigraphy and polysomnography devices (de Zambotti et al., 2019; Youngstedt 2003) and are broadly consistent with the expected night-to-night variability in these outcomes (Lolli et al., 2024b).

ELIGIBILITY:
Inclusion Criteria:

* Aspire Academy student-athlete (football)
* Healthy student-athletes currently injury-free and fully available for training and competition

Exclusion Criteria:

* Any participant not enrolled as Aspire Academy student-athlete
* Any Aspire Academy student-athlete currently facing any kind of sports injury

Ages: 13 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2025-09-21 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Time asleep | From enrollment to the end of treatment at 4 weeks.
  Time asleep, defined as 'the actual time that a person spends asleep excluding non-sleep-related activities in bed', tracked using actigraphy (ActiGraph GT9X Link monitors ) will represent the primary outcome measure in this investigation.

SECONDARY OUTCOMES:
Sleep onset latency | From enrollment to the end of treatment at 4 weeks.
  The time between lights out to the first epoch
Wake-after-sleep-onset | From enrollment to the end of treatment at 4 weeks.
  Periods of wakefulness occurring after defined sleep onset
Sleep efficiency | From enrolment to 4 weeks
  Time asleep divided by time in bed multiplied by 100
Sleep diary | From enrollment to the end of treatment at 4 weeks.
  Time someone went to bed; time someone thought fell asleep; time someone woke up.
Borg Ratings of perceived exertion (RPE) CR-100 scale (0-100) | From enrollment to the end of treatment at 4 weeks.
  Borg Category-Ratio 100 scale, a 0-100 scale used to measure perceived exertion during physical activity
High-speed running distance | From enrollment to the end of treatment at 4 weeks.
  Distance covered at high-speed running (>20 km/h) tracked using 10-Hz global positioning system.

CONTACTS AND LOCATIONS:
Locations (1):
- Aspire Academy, Football Performance and Science Department, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
The study will involve minors, and it will require additional approval from the Institutional Review Board given the Ministry of Public Health governance procedures in the State of Qatar.

REFERENCES:
- [Background] Deng C, Graz JC. Generating randomization schedules using SAS® programming. In N.W. Galwey (Ed.), Proceedings of the twenty-seventh annual SAS users group international conference (pp. 267-327). 2002.
- [Background] Senn S, Stevens L, Chaturvedi N. Repeated measures in clinical trials: simple strategies for analysis using summary measures. Stat Med. 2000 Mar 30;19(6):861-77. doi: 10.1002/(sici)1097-0258(20000330)19:63.0.co;2-f. PMID 10734289
- [Background] Zucker DR, Schmid CH, McIntosh MW, D'Agostino RB, Selker HP, Lau J. Combining single patient (N-of-1) trials to estimate population treatment effects and to evaluate individual patient responses to treatment. J Clin Epidemiol. 1997 Apr;50(4):401-10. doi: 10.1016/s0895-4356(96)00429-5. PMID 9179098
- [Background] Youngstedt SD. Ceiling and floor effects in sleep research. Sleep Med Rev. 2003 Aug;7(4):351-65. doi: 10.1053/smrv.2001.0239. PMID 14505601
- [Background] Walsh NP, Halson SL, Sargent C, Roach GD, Nedelec M, Gupta L, Leeder J, Fullagar HH, Coutts AJ, Edwards BJ, Pullinger SA, Robertson CM, Burniston JG, Lastella M, Le Meur Y, Hausswirth C, Bender AM, Grandner MA, Samuels CH. Sleep and the athlete: narrative review and 2021 expert consensus recommendations. Br J Sports Med. 2020 Nov 3:bjsports-2020-102025. doi: 10.1136/bjsports-2020-102025. Online ahead of print. PMID 33144349
- [Background] Viechtbauer W. Confidence intervals for the amount of heterogeneity in meta-analysis. Stat Med. 2007 Jan 15;26(1):37-52. doi: 10.1002/sim.2514. PMID 16463355
- [Background] Veroniki AA, Jackson D, Viechtbauer W, Bender R, Bowden J, Knapp G, Kuss O, Higgins JP, Langan D, Salanti G. Methods to estimate the between-study variance and its uncertainty in meta-analysis. Res Synth Methods. 2016 Mar;7(1):55-79. doi: 10.1002/jrsm.1164. Epub 2015 Sep 2. PMID 26332144
- [Background] Van Someren EJ, Cirelli C, Dijk DJ, Van Cauter E, Schwartz S, Chee MW. Disrupted Sleep: From Molecules to Cognition. J Neurosci. 2015 Oct 14;35(41):13889-95. doi: 10.1523/JNEUROSCI.2592-15.2015. PMID 26468189
- [Background] Tudor-Locke C, Barreira TV, Schuna JM Jr, Mire EF, Katzmarzyk PT. Fully automated waist-worn accelerometer algorithm for detecting children's sleep-period time separate from 24-h physical activity or sedentary behaviors. Appl Physiol Nutr Metab. 2014 Jan;39(1):53-7. doi: 10.1139/apnm-2013-0173. Epub 2013 Jun 26. PMID 24383507
- [Background] St-Onge MP, Mikic A, Pietrolungo CE. Effects of Diet on Sleep Quality. Adv Nutr. 2016 Sep 15;7(5):938-49. doi: 10.3945/an.116.012336. Print 2016 Sep. PMID 27633109
- [Background] Short MA, Arora T, Gradisar M, Taheri S, Carskadon MA. How Many Sleep Diary Entries Are Needed to Reliably Estimate Adolescent Sleep? Sleep. 2017 Mar 1;40(3):zsx006. doi: 10.1093/sleep/zsx006. PMID 28199718
- [Background] Shen T, Thackray AE, King JA, Alotaibi TF, Alanazi TM, Willis SA, Roberts MJ, Lolli L, Atkinson G, Stensel DJ. Are There Interindividual Responses of Cardiovascular Disease Risk Markers to Acute Exercise? A Replicate Crossover Trial. Med Sci Sports Exerc. 2024 Jan 1;56(1):63-72. doi: 10.1249/MSS.0000000000003283. Epub 2023 Aug 30. PMID 37703030
- [Background] Shamseer L, Sampson M, Bukutu C, Schmid CH, Nikles J, Tate R, Johnston BC, Zucker D, Shadish WR, Kravitz R, Guyatt G, Altman DG, Moher D, Vohra S; CENT Group. CONSORT extension for reporting N-of-1 trials (CENT) 2015: Explanation and elaboration. BMJ. 2015 May 14;350:h1793. doi: 10.1136/bmj.h1793. No abstract available. PMID 25976162
- [Background] Senn S. The analysis of continuous data from n-of-1 trials using paired cycles: a simple tutorial. Trials. 2024 Feb 16;25(1):128. doi: 10.1186/s13063-024-07964-7. PMID 38365817
- [Background] Senn S. Sample size considerations for n-of-1 trials. Stat Methods Med Res. 2019 Feb;28(2):372-383. doi: 10.1177/0962280217726801. Epub 2017 Sep 7. PMID 28882093
- [Background] Senn S. Mastering variation: variance components and personalised medicine. Stat Med. 2016 Mar 30;35(7):966-77. doi: 10.1002/sim.6739. Epub 2015 Sep 28. PMID 26415869
- [Background] Senn S. Suspended judgment n-of-1 trials. Control Clin Trials. 1993 Feb;14(1):1-5. doi: 10.1016/0197-2456(93)90045-f. No abstract available. PMID 8440091
- [Background] Senn S, Rolfe K, Julious SA. Investigating variability in patient response to treatment--a case study from a replicate cross-over study. Stat Methods Med Res. 2011 Dec;20(6):657-66. doi: 10.1177/0962280210379174. Epub 2010 Aug 25. PMID 20739334
- [Background] ROSE WC, WIXOM RL, LOCKHART HB, LAMBERT GF. The amino acid requirements of man. XV. The valine requirement; summary and final observations. J Biol Chem. 1955 Dec;217(2):987-95. No abstract available. PMID 13271458
- [Background] Reed DL, Sacco WP. Measuring Sleep Efficiency: What Should the Denominator Be? J Clin Sleep Med. 2016 Feb;12(2):263-6. doi: 10.5664/jcsm.5498. PMID 26194727
- [Background] Quante M, Kaplan ER, Cailler M, Rueschman M, Wang R, Weng J, Taveras EM, Redline S. Actigraphy-based sleep estimation in adolescents and adults: a comparison with polysomnography using two scoring algorithms. Nat Sci Sleep. 2018 Jan 18;10:13-20. doi: 10.2147/NSS.S151085. eCollection 2018. PMID 29403321
- [Background] Nikles J, Mitchell GK, Schluter P, Good P, Hardy J, Rowett D, Shelby-James T, Vohra S, Currow D. Aggregating single patient (n-of-1) trials in populations where recruitment and retention was difficult: the case of palliative care. J Clin Epidemiol. 2011 May;64(5):471-80. doi: 10.1016/j.jclinepi.2010.05.009. Epub 2010 Oct 8. PMID 20933365
- [Background] Mountjoy M, Sundgot-Borgen JK, Burke LM, Ackerman KE, Blauwet C, Constantini N, Lebrun C, Lundy B, Melin AK, Meyer NL, Sherman RT, Tenforde AS, Klungland Torstveit M, Budgett R. IOC consensus statement on relative energy deficiency in sport (RED-S): 2018 update. Br J Sports Med. 2018 Jun;52(11):687-697. doi: 10.1136/bjsports-2018-099193. No abstract available. PMID 29773536
- [Background] Merry TL, Ristow M. Do antioxidant supplements interfere with skeletal muscle adaptation to exercise training? J Physiol. 2016 Sep 15;594(18):5135-47. doi: 10.1113/JP270654. Epub 2016 Jan 18. PMID 26638792
- [Background] Maquet P. The role of sleep in learning and memory. Science. 2001 Nov 2;294(5544):1048-52. doi: 10.1126/science.1062856. PMID 11691982
- [Background] Lyon MR, Kapoor MP, Juneja LR. The effects of L-theanine (Suntheanine(R)) on objective sleep quality in boys with attention deficit hyperactivity disorder (ADHD): a randomized, double-blind, placebo-controlled clinical trial. Altern Med Rev. 2011 Dec;16(4):348-54. PMID 22214254
- [Background] Lolli L, Bonanno D, Lopez E, Di Salvo V. Night-to-night variability of objective sleep outcomes in youth Middle Eastern football players. Sleep Med. 2024 May;117:193-200. doi: 10.1016/j.sleep.2024.03.023. Epub 2024 Mar 19. PMID 38564918
- [Background] Lolli L, Cardinale M, Lopez E, Maasar MF, Marthinussen J, Bonanno D, Gregson W, Di Salvo V. An objective description of routine sleep habits in elite youth football players from the Middle-East. Sleep Med. 2021 Apr;80:96-99. doi: 10.1016/j.sleep.2021.01.029. Epub 2021 Jan 23. PMID 33588263
- [Background] Logan RW, McClung CA. Rhythms of life: circadian disruption and brain disorders across the lifespan. Nat Rev Neurosci. 2019 Jan;20(1):49-65. doi: 10.1038/s41583-018-0088-y. PMID 30459365
- [Background] Langan-Evans C, Hearris MA, Gallagher C, Long S, Thomas C, Moss AD, Cheung W, Howatson G, Morton JP. Nutritional Modulation of Sleep Latency, Duration, and Efficiency: A Randomized, Repeated-Measures, Double-Blind Deception Study. Med Sci Sports Exerc. 2023 Feb 1;55(2):289-300. doi: 10.1249/MSS.0000000000003040. Epub 2022 Sep 9. PMID 36094342
- [Background] Langan D, Higgins JPT, Jackson D, Bowden J, Veroniki AA, Kontopantelis E, Viechtbauer W, Simmonds M. A comparison of heterogeneity variance estimators in simulated random-effects meta-analyses. Res Synth Methods. 2019 Mar;10(1):83-98. doi: 10.1002/jrsm.1316. Epub 2018 Sep 6. PMID 30067315
- [Background] Lakens D. Sample size justification. Collabra Psychol. 2022;8(1):33267.
- [Background] Knutson KL, Rathouz PJ, Yan LL, Liu K, Lauderdale DS. Intra-individual daily and yearly variability in actigraphically recorded sleep measures: the CARDIA study. Sleep. 2007 Jun;30(6):793-6. doi: 10.1093/sleep/30.6.793. PMID 17580601
- [Background] Johnston RD, Hewitt A, Duthie G. Validity of Real-Time Ultra-wideband Global Navigation Satellite System Data Generated by a Wearable Microtechnology Unit. J Strength Cond Res. 2020 Jul;34(7):2071-2075. doi: 10.1519/JSC.0000000000003059. PMID 32598123
- [Background] IntHout J, Ioannidis JP, Rovers MM, Goeman JJ. Plea for routinely presenting prediction intervals in meta-analysis. BMJ Open. 2016 Jul 12;6(7):e010247. doi: 10.1136/bmjopen-2015-010247. PMID 27406637
- [Background] IntHout J, Ioannidis JP, Borm GF. The Hartung-Knapp-Sidik-Jonkman method for random effects meta-analysis is straightforward and considerably outperforms the standard DerSimonian-Laird method. BMC Med Res Methodol. 2014 Feb 18;14:25. doi: 10.1186/1471-2288-14-25. PMID 24548571
- [Background] Hannon MP, Parker LJF, Carney DJ, McKeown J, Speakman JR, Hambly C, Drust B, Unnithan VB, Close GL, Morton JP. Energy Requirements of Male Academy Soccer Players from the English Premier League. Med Sci Sports Exerc. 2021 Jan;53(1):200-210. doi: 10.1249/MSS.0000000000002443. PMID 32701871
- [Background] Gonzalez JT, Lolli L, Veasey RC, Rumbold PLS, Betts JA, Atkinson G, Stevenson EJ. Are there interindividual differences in the reactive hypoglycaemia response to breakfast? A replicate crossover trial. Eur J Nutr. 2024 Dec;63(8):2897-2909. doi: 10.1007/s00394-024-03467-y. Epub 2024 Sep 4. PMID 39231870
- [Background] Goltz FR, Thackray AE, Atkinson G, Lolli L, King JA, Dorling JL, Dowejko M, Mastana S, Stensel DJ. True Interindividual Variability Exists in Postprandial Appetite Responses in Healthy Men But Is Not Moderated by the FTO Genotype. J Nutr. 2019 Jul 1;149(7):1159-1169. doi: 10.1093/jn/nxz062. PMID 31132105
- [Background] Goltz FR, Thackray AE, King JA, Dorling JL, Atkinson G, Stensel DJ. Interindividual Responses of Appetite to Acute Exercise: A Replicated Crossover Study. Med Sci Sports Exerc. 2018 Apr;50(4):758-768. doi: 10.1249/MSS.0000000000001504. PMID 29240652
- [Background] Garlick PJ. The nature of human hazards associated with excessive intake of amino acids. J Nutr. 2004 Jun;134(6 Suppl):1633S-1639S; discussion 1664S-1666S, 1667S-1672S. doi: 10.1093/jn/134.6.1633S. PMID 15173443
- [Background] Fox JL, Scanlan AT, Stanton R, Sargent C. Insufficient Sleep in Young Athletes? Causes, Consequences, and Potential Treatments. Sports Med. 2020 Mar;50(3):461-470. doi: 10.1007/s40279-019-01220-8. PMID 31679145
- [Background] Fernstrom JD. Effects and side effects associated with the non-nutritional use of tryptophan by humans. J Nutr. 2012 Dec;142(12):2236S-2244S. doi: 10.3945/jn.111.157065. Epub 2012 Oct 17. PMID 23077193
- [Background] Elango R. Tolerable Upper Intake Level for Individual Amino Acids in Humans: A Narrative Review of Recent Clinical Studies. Adv Nutr. 2023 Jul;14(4):885-894. doi: 10.1016/j.advnut.2023.04.004. Epub 2023 Apr 14. PMID 37062432
- [Background] Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. BMJ. 2019 Jul 31;366:l4378. doi: 10.1136/bmj.l4378. PMID 31366597
- [Background] Di Salvo V, Gregson W, Atkinson G, Tordoff P, Drust B. Analysis of high intensity activity in Premier League soccer. Int J Sports Med. 2009 Mar;30(3):205-12. doi: 10.1055/s-0028-1105950. Epub 2009 Feb 12. PMID 19214939
- [Background] Coates S, Taubel J, Lorch U. Practical risk management in early phase clinical trials. Eur J Clin Pharmacol. 2019 Apr;75(4):483-496. doi: 10.1007/s00228-018-02607-8. Epub 2018 Dec 19. PMID 30569285
- [Background] Cynober L, Bier DM, Kadowaki M, Morris SM Jr, Elango R, Smriga M. Proposals for Upper Limits of Safe Intake for Arginine and Tryptophan in Young Adults and an Upper Limit of Safe Intake for Leucine in the Elderly. J Nutr. 2016 Dec;146(12):2652S-2654S. doi: 10.3945/jn.115.228478. Epub 2016 Nov 9. PMID 27934658
- [Background] de Zambotti M, Cellini N, Goldstone A, Colrain IM, Baker FC. Wearable Sleep Technology in Clinical and Research Settings. Med Sci Sports Exerc. 2019 Jul;51(7):1538-1557. doi: 10.1249/MSS.0000000000001947. PMID 30789439
- [Background] Covassin N, Singh P, McCrady-Spitzer SK, St Louis EK, Calvin AD, Levine JA, Somers VK. Effects of Experimental Sleep Restriction on Energy Intake, Energy Expenditure, and Visceral Obesity. J Am Coll Cardiol. 2022 Apr 5;79(13):1254-1265. doi: 10.1016/j.jacc.2022.01.038. PMID 35361348
- [Background] Chatters R, Hawksworth O, Julious S, Cook A. The development of a set of key points to aid clinicians and researchers in designing and conducting n-of-1 trials. Trials. 2024 Jul 11;25(1):473. doi: 10.1186/s13063-024-08261-z. PMID 38992786
- [Background] Bruni O, Ferri R, Miano S, Verrillo E. L -5-Hydroxytryptophan treatment of sleep terrors in children. Eur J Pediatr. 2004 Jul;163(7):402-7. doi: 10.1007/s00431-004-1444-7. Epub 2004 May 14. PMID 15146330
- [Background] Borenstein M. Avoiding common mistakes in meta-analysis: Understanding the distinct roles of Q, I-squared, tau-squared, and the prediction interval in reporting heterogeneity. Res Synth Methods. 2024 Mar;15(2):354-368. doi: 10.1002/jrsm.1678. Epub 2023 Nov 8. PMID 37940120
- [Background] Barrett JR, Tracy DK, Giaroli G. To sleep or not to sleep: a systematic review of the literature of pharmacological treatments of insomnia in children and adolescents with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2013 Dec;23(10):640-7. doi: 10.1089/cap.2013.0059. Epub 2013 Nov 21. PMID 24261659
- [Background] Bacchetti P. Current sample size conventions: flaws, harms, and alternatives. BMC Med. 2010 Mar 22;8:17. doi: 10.1186/1741-7015-8-17. PMID 20307281
- [Background] Atkinson G, Batterham AM. True and false interindividual differences in the physiological response to an intervention. Exp Physiol. 2015 Jun;100(6):577-88. doi: 10.1113/EP085070. Epub 2015 May 13. PMID 25823596
- [Background] Atkinson G, Williamson P, Batterham AM. Issues in the determination of 'responders' and 'non-responders' in physiological research. Exp Physiol. 2019 Aug;104(8):1215-1225. doi: 10.1113/EP087712. Epub 2019 Jun 9. PMID 31116468